CLINICAL TRIAL: NCT06310980
Title: Pilot Study in Order to Verify the Effect of the Use of a Smartpen Coordinated With a Continuous Glucose Sensor by a Dedicated App, in a Group of Adolescents in Not Good Control: Sensor Augmented Smartpen.
Brief Title: Pilot Study to Verify Effect of Smartpen Coordinated With Glucose Sensor.
Acronym: SMARTPEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Giulio Frontino (Other)
Responsible Party: Sponsor-Investigator, Giulio Frontino, sub investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMARTPEN
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- smartpen (Experimental): patients treated by smartpen, glucose sensor and connected by a digital application
  Interventions: Device: smartpen

INTERVENTIONS:
Device: smartpen — use of a smartpen connected with glucose sensor by an digital application

SUMMARY:
The Aim of this interventional study in to assess the effect of the use of a smartpen connected by an APP to continuous glucose sensors in a cohort of diabetic adolescents in not good metabolic control.

Primary endpoint: time in range Secondary endpoints: other glucometrics, Hba1c, treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12 - 18 years
2. A clinical diagnosis of diabetes type 1 as determined by investigator for at least 12 months.
3. HbA1c >7.5% (DCA)
4. Subject is on multiple daily injection therapy (3 or more insulin injections per day one of which is a long acting insulin injection), is currently using or is willing to use insulin pens and pen cartridges and are not willing to use an insulin pump or AHCL system
5. Subject is currently using a CGM or is willing to use the Guardian 4 system during the study.
6. Subject and parents agree to comply with the study protocol requirements
7. Subject and parents provide their signature on the Informed Consent Form

Exclusion Criteria:

1. Subject is unwilling or unable to use insulin pen(s).
2. Subject is in plans to use or is already using an insulin pump.
3. Subject is currently using a non-Medtronic standalone CGM system and unwilling to use only the Guardian 4 system during the study.
4. Subject has any unresolved adverse skin condition in the area of device placement (e.g. psoriasis, rash, Staphylococcus infection).
5. Subject is actively participating in or plans to enroll in an investigational study (e.g. drug or device), other than this study, wherein they have received treatment from an investigational drug or device.
6. Subject has a positive urine pregnancy test at time of screening.
7. Subject is unwilling to participate in study procedures.
8. Subject is directly involved in the study as research staff.
9. Subject with poorly controlled thyroid or celiac disease.
10. Subject with any risk of exposure to MRI equipment, diathermy devices or other devices capable of generating strong magnetic fields

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Time in range | 3 months
  Percentage of the time spent by 70-180 mg/dl

SECONDARY OUTCOMES:
time below range | 3 months
  percentage of time < 70 mg/dl
time above range | 3 months
  percentage of time spent > 180 mg/dl
coefficient of variation (CV) | 3 months
  percentage of variation of glicaemic values
HbA1c | 3 months
  percentage of glicated haemoglobin
ITSRQ | end of the study
  questionnaire on patient's satisfaction about the use of insulin device
DIDS | 3 months
  questionnaire on patient's satisfaction about the use of insulin device

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Bonfanti, M.D., Principal Investigator — IRCCS San Raffaele